CLINICAL TRIAL: NCT07388108
Title: Atrial Electromechanical Alteration as a Predictor of Arrhythmias in the Postoperative Period After Cardiovascular Surgery
Brief Title: Atrial Dyssynchrony to Predict Arrhythmias in the Postoperative Setting of Cardiovascular Surgery.
Acronym: SAD-POAF
Status: Recruiting | Type: Observational
Sponsor: School of Medicine. National University of Cuyo (Other)
Responsible Party: Principal Investigator, Francisco Javier Sánchez, MD; PhD, School of Medicine. National University of Cuyo
Other Study IDs: 003. 03/10/2023.
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Postoperative Complications
Keywords: Atrial fibrillation; Atrial strain; Cardiovascular surgery; Echocardiography
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Atrial dyssynchrony — To determine interatrial dyssynchrony, an adaptation of the echocardiographic atrial strain will be made so that both atria can be evaluated simultaneously. This new evaluation, OMEGA (ω) will yield the time to maximum deformation of the lateral segments of the right atrium and the lateral segments of the left atrium.
  Additionally, total atrial deformation will be evaluated via bi-atrial strain analysis. We will then measure the maximum deformation time-from P-wave onset to the maximum negative strain deflection-to assess its relationship with atrial contraction strain.

SUMMARY:
This study aims to improve the prediction for developing arrhythmias in the postoperative period of cardiovascular surgery by using non-invasive echocardiographic techniques that are sensitive to detect inter and intra-atrial dyssynchrony. The main question it aims to answer is:

Do patients with atrial dyssynchrony are at increased risk of developing arrhythmias in the postoperative period of cardiovascular surgery?

Patients admitted to the protocol will undergo an echocardiogram with atrial strain before surgery to determine the presence or absence of intra- and inter-atrial dyssynchrony and will be followed during hospitalization to assess the occurrence of atrial fibrillation in the postoperative period.

DETAILED DESCRIPTION:
The overall objective is to improve the prediction of the risk of developing arrhythmias in the postoperative period with non-invasive techniques that are sensitive to detect inter- and intra-atrial dysrhythmias.

Specific objectives

1. To describe the alterations in left and right atrial deformation by strain method to identify intra- and inter-atrial activation dyssynchrony.
2. To determine that dyssynchrony predicts a higher incidence of atrial fibrillation in the postoperative period after cardiovascular surgery.
3. To evaluate whether novel atrial function analysis techniques, such as left atrial ejection fraction assessed via 3D echocardiography, are associated with a higher incidence of postoperative atrial fibrillation.

All patients will undergo a full Doppler echocardiogram with two-dimensional atrial Strain determination with speckle tracking, using an Philips EPIC CVx series echocardiogram machine with S5-1 and X5-1 probes. The images will be obtained in left lateral decubitus. In forced expiration, 3 consecutive beats will be recorded and digitally saved for later analysis in the 4 and 2 chamber views. Both atria must be visualized so that neither atrial wall are lost in the evaluation. Echocardiographic measurements will focus primarily on the indexed left atrial volume obtained by averaging the values obtained in 2 and 4 chambers by the multiple disc method. In these views, the left ventricular ejection fraction will be obtained by the Simpson biplane method. The left atrium will be further subdivided into basal, medial and atrial roof segments, resulting in a total of 12 segments, 6 of which can be observed in the four-chamber view and 6 in the two-chamber view. The right atrium will be divided similarly but will contribute a mere three additional segments to the total (for a total of 15 segments), as the right septal segments were previously regarded as part of the left atrium. The time to maximum deflection, defined as the interval between the onset of the P wave on the electrocardiogram and the maximum deflection of the atrial contraction determined by strain rate, will be measured for each of the 15 atrial segments previously described. To determine interatrial synchrony, an adaptation of the atrial strain will be made so that both atria can be evaluated simultaneously. This new evaluation, which we have designated "OMEGA" (ω) due to its resemblance to the shape of the strain image, will yield the time to maximum deformation of the lateral segments of the right atrium and the lateral segments of the left atrium. Consequently, the difference in activation timing between the lateral segments of the right and left atria will determine the presence of an activation delta between the walls.

A comprehensive analysis of atrial deformation using left and right atrial strain will also be performed. Subsequently, the time-to-peak deformation will be measured from the onset of the P-wave to the peak negative atrial strain deflection, which correlates with atrial contractile strain. Activation time differences derived from this methodology will also be measured to provide an additional assessment of the interatrial activation delay (delta).

Patients will be followed during hospitalization with continuous electrocardiographic monitoring for the first 5 days after surgery to detect the incidence of atrial fibrillation. Patients will undergo telephonic follow-up at 28 and 365 days post-intervention, utilizing a targeted interview to evaluate for the onset of supraventricular arrhythmias.

Study data will be collected and managed using REDCap electronic data capture tools hosted at Faculty of Medicine, National University of Cuyo to a protocol designed specifically for this study.

The sample size calculation is performed according to Schoenfeld's method for Cox models. To detect a hazard ratio of 2.5 for atrial fibrillation events based on the presence or absence of interatrial dyssynchrony-estimating a cumulative event rate of 0.38 in the dyssynchronous group and 0.18 in the synchronous group, with a 0.44 proportion of dyssynchronous patients-and assuming a two-sided alpha level of 0.05 and 80% power, a total sample of 138 patients is determined.

Statistical analysis results are reported as mean (SD), median (p25-p75) or frequency (%). Comparisons between groups were performed with the Student t test or chi-squared analysis. The association between clinical variables and the study end-points was evaluated using survival analysis methodology (Cox regression models). The Kaplan-Meier method was used to estimate the cumulative probability of PAF detection and stroke recurrence in both groups, and comparisons were made by the log-rank test. Significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with criteria for non-mitral cardiovascular surgery, in sinus rhythm, and who gave informed consent to participate in the study.
* Absence of atrial fibrillation upon hospital admission for surgery.

Exclusion Criteria:

* Surgery of the mitral or tricuspid valve.
* History of previous atrial fibrillation.
* History of congenital heart disease or cardiac tumors.
* Emergency surgery of the heart
* Pour echocardiographic window

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of coronary artery disease, aortic stenosis or a combination of both pathologies, with indication for cardiovascular surgery according to the Guidelines for Cardiovascular Surgery of the European Society of Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperatory atrial fibrillation | From the end of surgery through hospital discharge, an average of 6 days.
  Arrhythmic episodes of at least 30 seconds duration will be considered postoperative atrial fibrillation when detected on continuous monitoring or when detected on a ward ECG, if the patient reported symptoms or required medical intervention.

SECONDARY OUTCOMES:
Atrial Fibrillation at 28 and 365 Days | From surgery through Day 28 and Day 365
  Telephone follow-ups will be conducted with all patients at 28 and 365 days post-surgery. A brief interview will be administered to screen for the occurrence of arrhythmias during this period. Patients reporting a positive history will be scheduled for an on-site visit to request diagnostic tests documenting the arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Diez, PhD, Study Director — National University of Cuyo
Locations (1):
- Clínica de Cuyo, Mendoza, Mendozz, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The data dictionary of analyzed variables and the corresponding statistical analysis will be available upon formal request by email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The information will be available three months following the completion of patient enrollment and for a duration of five years thereafter.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Background] Sánchez FJ, Gonzalez VA, Farrando M, Baigorria Jayat AO, Segovia-Roldan M, García-Mendívil L, Ordovás L, Prado NJ, Pueyo E, Diez ER. Atrial Dyssynchrony Measured by Strain Echocardiography as a Marker of Proarrhythmic Remodeling and Oxidative Stress in Cardiac Surgery Patients. Oxid Med Cell Longev. 2020:8895078.
- [Background] Badano, L.P.; Kolias, T.J.; Muraru, D.; Abraham, T.P.; Aurigemma, G.; Edvardsen, T.; D'Hooge, J.; Donal, E.; Fraser, A.G.; Marwick, T.; et al. Standardization of left atrial, right ventricular, and right atrial deformation imaging using two-dimensional speckle tracking echocardiography: A consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. Eur. Heart J. Cardiovasc. Imaging 2018, 19, 591-600, doi:10.1093/ehjci/jey042.
- [Background] Aksu, U.; Kalkan, K.; Gulcu, O.; Aksakal, E.; Öztürk, M.; Topcu, S. The role of the right atrium in development of postoperative atrial fibrillation: A speckle tracking echocardiography study. J. Clin. Ultrasound 2019, 47, 470-476, doi:10.1002/jcu.22736.
- [Background] Müller, P.M.; Hars, C.; Schiedat, F.; Osche, L.I.B.; Gotzmann, M.; Strauch, J.; Dietrich, J.W.; Vogt, M.; Tannapfel, A.; Deneke, T.; et al. Correlation Between Total Atrial Conduction Time Estimated via Tissue Doppler Imaging ( PA-TDI Interval ), Structural Atrial Remodeling and New-Onset of Atrial Fibrillation. J. Cardiovasc. Electrophysiol. 2013, 24, 626-631, doi:10.1111/jce.12084
- [Background] Merckx, K.L.; Vos, C.B. De; Palmans, A.; Habets, J.; Tieleman, R.G. Atrial Activation Time Determined by Transthoracic Doppler Tissue Imaging Can Be Used as an Estimate of the Total Duration of Atrial Electrical Activation. 940-944, doi:10.1016/j.echo.2005.03.022.
- [Background] Xu, C.; Chen, K.; Yu, F.; Wang, Q.; Su, H.; Yang, D.; Xu, J.; Yan, J. Atrial Dyssynchrony: A New Predictor for Atrial High-Rate Episodes in Patients with Cardiac Resynchronization Therapy. Cardiol. 2019, 144, 18-26, doi:10.1159/000502541.
- [Background] Ciuffo, L.; Tao, S.; Gucuk Ipek, E.; Zghaib, T.; Balouch, M.; Lima, J.A.C.; Nazarian, S.; Spragg, D.D.; Marine, J.E.; Berger, R.D.; et al. Intra-Atrial Dyssynchrony During Sinus Rhythm Predicts Recurrence After the First Catheter Ablation for Atrial Fibrillation. JACC Cardiovasc. Imaging 2019, 12, 310-319, doi:10.1016/j.jcmg.2017.11.028.
- [Background] . Pathan, F.; D'Elia, N.; Nolan, M.T.; Marwick, T.H.; Negishi, K. Normal Ranges of Left Atrial Strain by Speckle-Tracking Echocardiography: A Systematic Review and Meta-Analysis. J. Am. Soc. Echocardiogr. 2017, 30, 59-70.e8, doi:10.1016/j.echo.2016.09.007.
- [Background] Swartz, M.F.; Fink, G.W.; Sarwar, M.F.; Hicks, G.L.; Yu, Y.; Hu, R.; Lutz, C.J.; Taffet, S.M.; Jalife, J. Elevated pre-operative serum peptides for collagen i and III synthesis result in post-surgical atrial fibrillation. J. Am. Coll. Cardiol. 2012, 60, 1799-1806, doi:10.1016/j.jacc.2012.06.048.
- [Background] Lacalzada-Almeida, J.; Izquierdo-Gómez, M.M.; Belleyo-Belkasem, C.; Barrio-Martínez, P.; GarcíaNiebla, J.; Elosua, R.; Jiménez-Sosa, A.; Escobar-Robledo, L.A.; Bayés de Luna, A. Interatrial block and atrial remodeling assessed using speckle tracking echocardiography. BMC Cardiovasc. Disord. 2018, 18, 1-9, doi:10.1186/s12872-018-0776-6.
- [Background] Hatam, N.; Aljalloud, A.; Mischke, K.; Karfis, E.A.; Autschbach, R.; Hoffmann, R.; Goetzenich, A. Interatrial conduction disturbance in postoperative atrial fibrillation: A comparative study of P-wave dispersion and Doppler myocardial imaging in cardiac surgery. J. Cardiothorac. Surg. 2014, 9, 1-9, doi:10.1186/1749-8090-9-114
- [Background] Osranek, M.; Kaniz, F.; Fatema, Q.; Al-Saileek, A.; Barnes, M.E.; Bailey, K.R. Left Atrial Volume Predicts the Risk of Atrial Fibrillation After Cardiac Surgery A Prospective Study. J. Am. Coll. Cardiol. 2006, 48, doi:10.1016/j.jacc.2006.03.054.
- [Background] Liberale, L.; Montecucco, F.; Tardif, J.C.; Libby, P.; Camici, G.G. Inflamm-ageing: the role of inflammation in age- dependent cardiovascular disease. Eur. Heart J. 2020, 41, 2974-2982, doi:10.1093/eurheartj/ehz961.
- [Background] . Zakkar, M.; Ascione, R.; James, A.F.; Angelini, G.D.; Suleiman, M.S. Inflammation, oxidative stress and postoperative atrial fibrillation in cardiac surgery. Pharmacol. Ther. 2015, 154, 13-20, doi:10.1016/j.pharmthera.2015.06.009.
- [Background] Maesen, B.; Nijs, J.; Maessen, J.; Allessie, M.; Schotten, U. Post-operative atrial fibrillation: A maze of mechanisms. Europace 2012, 14, 159-174, doi:10.1093/europace/eur208.
- [Background] Akintoye, E.; Sellke, F.; Marchioli, R.; Tavazzi, L.; Mozaffarian, D. Factors associated with postoperative atrial fibrillation and other adverse events after cardiac surgery. J. Thorac. Cardiovasc. Surg. 2018, 155, 242-251.e10, doi:10.1016/j.jtcvs.2017.07.063.
- [Background] . Steinberg, B.A.; Zhao, Y.; He, X.; Hernandez, A.F.; Fullerton, D.A.; Thomas, K.L.; Mills, R.; Klaskala, W.; Peterson, E.D.; Piccini, J.P. Quality and Outcomes Management of Postoperative Atrial Fibrillation and Subsequent Outcomes in Contemporary Patients Undergoing Cardiac Surgery : Insights From the Society of Thoracic Surgeons CAPS-Care Atrial Fibrillation Registry. 2014, 13, 7-13, doi:10.1002/clc.22230.
- [Background] Júnior, F.P.; Filho, G.F.T.; Sant'anna, J.R.M.; Py, P.M.; Prates, P.R.; Nesralla, I.A.; Kalil, R.A. Idade avançada e incidência de fibrilação atrial em pós-operatório de troca valvar aórtica. Brazilian J. Cardiovasc. Surg. 2014, 29, 45-50, doi:10.5935/1678-9741.20140010.